CLINICAL TRIAL: NCT03275909
Title: Integrated Psychological Therapy (IPT) + Emotional Management Therapy (EMT) in Chronic Schizophrenia: Study Protocol for a Randomized Controlled Trial
Brief Title: Integrated Psychological Therapy for Chronic Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Karmele Salaberria Irizar, Phd.-Lecturer, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI2011-27590
Record Dates: First submitted 2017-07-10; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Chronic Schizophrenia
Keywords: Chronic schizophrenia; Emotional Management Therapy; Integrated Psychological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study procedure (Experimental): An experimental group the psychological treatment includes 50 sessions of integrated psychological therapy (IPT) (focused on attentional skills training, social perception skills training, verbal communication skills, social skills training, interpersonal problems solving skills) and 10 sessions of specific emotional management therapy (EMT), designed for this research and based on the contents developed by Hodel, Kern and Brenner.
  Interventions: Behavioral: Integrated Psychological Therapy
- Treatment as usual (No Intervention): The treatment as usual is pharmacological treatment and activities in a Day Care Center.

INTERVENTIONS:
Behavioral: Integrated Psychological Therapy — The psychological treatment includes 50 sessions of integrated psychological therapy focused on attentional skills, social perception skills, verbal communication skills, social skills and interpersonal problems solving skills and 10 sessions of specific emotional management therapy , designed for this research. and based on the contents developed by Hodel, Kern and Brenner
  Other Names: Emotional Management Therapy
  Arms: Study procedure

SUMMARY:
Background: The chronic phase of schizophrenia (CS) that extremely affects the way people think, feel and act, underlines the need for effective interventions in patients affected by this disorder. The Integrated Psychological Therapy appears in clinical practice guidelines as the reference therapy in the treatment of this type of patients. In this paper authors propose to include in this program a new module focused on Emotional Management Therapy in order to reinforce its effectiveness. The aim of this study is to describe the design of a study protocol for a randomized controlled trial in which the objective is to assess the efficacy of this modified IPT program in patients with CS compared to treatment as usual (pharmacological treatment and social and leisure activities in a Day Care Center).

Methods/design: This is a randomized study with pre and post-treatment assessment and with a 6- and 12-month follow-up. Patients are to be randomly assigned to one of two treatments: (1) a experimental group: integrated psychological therapy in conjunction with emotional management therapy (IPT+EMT), composed of 2-hour biweekly 60 group sessions for 32 weeks, in addition to the treatment as usual (TAU), or (2) a control group (treatment as usual). Participants in both groups will be evaluated at baseline (pre-treatment) and at post-treatment after 8 months. The primary outcome will be that patients in the experimental group will show a greater improvement over participants in the control group in reducing symptoms and increasing emotional abilities, as well as in improving their quality of life. The secondary outcome will be that these results will maintain at the 6- and 12-month follow-up in the experimental group.

DETAILED DESCRIPTION:
Background: The chronic phase of schizophrenia (CS) that extremely affects the way people think, feel and act, underlines the need for effective interventions in patients affected by this disorder. The Integrated Psychological Therapy (IPT) appears in clinical practice guidelines as the reference therapy in the treatment of this type of patients. In this paper authors propose to include in this program a new module focused on Emotional Management Therapy (EMT) in order to reinforce its effectiveness. The aim of this study is to describe the design of a study protocol for a randomized controlled trial in which the objective is to assess the efficacy of this modified IPT program in patients with CS compared to treatment as usual (pharmacological treatment and social and leisure activities in a Day Care Center).

Methods/design: This is a randomized study with pre and post-treatment assessment and with a 6- and 12-month follow-up. Patients are to be randomly assigned to one of two treatments: (1) a experimental group: integrated psychological therapy in conjunction with emotional management therapy (IPT+EMT), composed of 2-hour biweekly 60 group sessions for 32 weeks, in addition to the treatment as usual (TAU), or (2) a control group (treatment as usual). Participants in both groups will be evaluated at baseline (pre-treatment) and at post-treatment after 8 months. The primary outcome will be that patients in the experimental group will show a greater improvement over participants in the control group in reducing symptoms and increasing emotional abilities, as well as in improving their quality of life. The secondary outcome will be that these results will maintain at the 6- and 12-month follow-up in the experimental group.

Discussion: This study provides the description of a clinical trial based on specific psychological intervention (IPT+EMT) for patients with chronic schizophrenia, aiming to improve lasting clinical and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Having ≥ 5 years since disease onset and aged between 25 and 65 years.
2. Being in a stable phase of the illness and under psychopharmacological treatment.
3. Having negative or attenuated positive symptoms.
4. Failing to achieve premorbid functioning in terms of education, work and/or social life.
5. Agreeing to participate in the study and giving written informed consent.

Exclusion Criteria:

* 1. Presenting organic brain pathology. 2. Presenting intellectual developmental disorder according to DSM-5 criteria.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Frankfurt Complaint Questionnaire (FBF-3) | Pretreatment-Posttreatment (8months)-1 month-3 months-6 months-12 months follow-up
  (Assessing change)This is a self-report test composed of 98 items measuring the presence of the "basic" symptoms of schizophrenia. These are subjectively experienced disturbances at different domains including perception, thought, processing, language and attention that it could be the neurobiological features of schizophrenia. It contains 10 subscales and 4 factors. We will use a validated version for the Spanish population, in which Cronbach's alpha was above .95 and the test-retest reliability was above .60

SECONDARY OUTCOMES:
Screen for Cognitive Impairment in Psychiatry (SCIP) | Pretreatment-Posttreatment (8 months)-1 month-3 months-6 months-12 months follow-up
  (Assessing change)This test assesses cognitive impairment through five areas: immediate and delayed verbal learning, working memory, verbal fluency and information processing speed. It is used for identifying cognitive impairment. The test-retest reliability ranged from 74 to 90 and Cronbach's alpha was 73.
Wechsler Adult Intelligence Scale-Third Edition (WAIS-III) | Pretreatment-Posttreatment (8 months)-1 month-3 months-6 months-12 months follow-up
  (Assessing change)Short forms of this scale have been designed for patients with schizophrenia . It assess cognitive functioning. Scores on these short forms are correlated (0.91) with the overall intelligence quotient (IQ) of the full scale in clinical patients.
Wisconsin Card Sorting Test (WCST) | Pretreatment-Posttreatment (8 months)-1 month-3 months-6 months-12 months follow-up
  (Assessing change)This test assesses attention span, planning and execution, and hence is considered a valid measure of executive function. We used the version of the test standardised and benchmarked for the Spanish population by TEA Editions.
Social Functioning Scale (SFS) | Pretreatment-Posttreatment-1 month (8 months)-3 months-6 months-12 months follow-up
  (Assessing change)We will use the short version of the scale, validated in a Spanish clinical sample, with a Cronbach's alpha of 0.76.
Lancashire Quality of Life Profile (LQoLP) | Pretreatment-Posttreatment (8 months)-1 month-3 months-6 months-12 months follow-up
  (Assessing change)This instrument assesses patient satisfaction with various aspects of their life, work, leisure time, religion, finances, living situation, safety, family relations, social relations, and health, as well as global wellbeing and self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Karmele Salaberria, Ph.D, Principal Investigator — Lecturer of School of Psychology

IPD SHARING:
Plan to Share IPD: Yes
to share the study protocol and the clinical study report
Supporting Information: Study Protocol, CSR
Time Frame: 2011/2017
Access Criteria: Researchers

DOCUMENTS (3):
  • Informed Consent Form (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03275909/ICF_000.pdf
  • Statistical Analysis Plan (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03275909/SAP_001.pdf
  • Study Protocol (2013-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03275909/Prot_002.pdf